CLINICAL TRIAL: NCT03473457
Title: The Prospective, Multi-center And Single-arm Clinical Study of Chimeric Antigen Receptor T(CAR-T) Cells Therapy in Relapsed/Refractory Acute Myeloid Leukemia
Brief Title: CAR-T Cells Therapy in Relapsed/Refractory Acute Myeloid Leukemia
Acronym: AML
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The therapeutic effect was not as expected
Sponsor: Zhujiang Hospital (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); The Third Affiliated Hospital of Southern Medical University (Other Government); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-XYNK-002
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Relapsed/Refractory Acute Myeloid Leukemia(AML)
Keywords: CD38-CART; CD33-CART; CD56-CART; CD123-CART; CD117-CART; CD133-CART; CD34-CART; Mucl-CART
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CART therapy in Acute myeloid leukemia (Experimental): In order to assess the safety and validity of using CAR-T therapy refractory/relapsed acute myeloid leukemia（AML）patients with one kind of CD38-CART/CD33-CART/CD56-CART/CD123-CART/CD117-CART/CD133-CART/CD34-CART/Mucl-CART,subjects will receive 10^6-10^7/Kg transduced CAR T cells at one time.
  Interventions: Biological: CART therapy in Acute myeloid leukemia(AML)

INTERVENTIONS:
Biological: CART therapy in Acute myeloid leukemia(AML) — one kind of CD38-CART/CD33-CART/CD56-CART/CD123-CART/CD117-CART/CD133-CART/CD34-CART/Mucl-CART therapy in Acute myeloid leukemia(AML)

SUMMARY:
Acute myeloid leukemia (AML) is a group of genetically highly heterogeneous malignant disease . The disease is the most common type of adult acute leukemia. Overall survival (OS) was less than 50% in 5 years. Chimeric Antigen Receptor-transduced T cell (CAR-T) therapy is one of revolutionary targeted immunotherapy. The efficacy of CAR-T cells for the treatment of acute B lymphocytic leukemia has been widely recognized, although it start late, several clinical trials have been register in ClinicalTrials.gov.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a group of genetically highly heterogeneous malignant disease ,its' character is immature myeloid protocel abnormal differentiation and proliferation in the bone marrow. The disease is the most common type of adult acute leukemia, Overall survival (OS) was less than 50% in 5 years. Chimeric Antigen Receptor-transduced T cell (CAR-T) therapy is one of revolutionary targeted immunotherapy.

CAR - T cells are taken in the form of genetic modification, and specific identified target antigen monoclonal antibody of single variable region (scFv) expression in T cell surface, and coupled with the activation of intracellular proliferation signal domain.When scFv recognizes antigens expressed in malignant cells, it stimulates the activation signal of downstream T cells and produces specific killing effects. CAR-T therapy is one of revolutionary targeted immunotherapy.The efficacy of CAR-T cells for the treatment of acute B lymphocytic leukemia has been widely recognized, although it start late, several clinical trials have been register in ClinicalTrials.gov.

The cluster of differentiation (CD) antigen serves as the target for identification and research in the immuno-phenotype detection of cells.As the surface markers of immune typing, CD molecules can be used as cell identification for expression types and levels on the cell surface.Cell surface of AML has a specific type of CD molecule expression,such as cluster of differentiation antigen 33(CD33),cluster of differentiation 38(CD38),cluster of differentiation 56 (CD56), cluster of differentiation 123(CD123), cluster of differentiation 117(CD117), cluster of differentiation 133(CD133), cluster of differentiation 34(CD34) and Mucl.Therefore, it provides some good targets for the immunotherapy of CAR T cells.In AML cells and mouse model,some studies have confirmed anti-CD33 CAR-T and anti-CD123 CAR-T with good similar lethality, but the toxicity of CAR-T to myeloid hematopoietic stem/progenitor cells and mononuclear cells is widespread.In comparison,CD123 CAR-T Off-target effects slighter than CD33 CAR-T.

In order to lay a foundation for the application of relapsed/refractory AML patients with CAR-T therapy，objects are refractory/ relapsed patients with AML,and plans to into the group of the number of cases in 50 cases.The main content is safety, efficacy and feasibility analysis of the CAR-T cells （single CAR-T or double CAR-T cells with CD33,CD38,CD56,CD123,CD117,CD133,CD34 or Mucl ) in the treatment of refractory/relapsed AML.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed/Refractory AML patients
2. Positive for any of CD33, CD38, CD56, CD117, CD123, CD34, or Muc1.(cytology, genetic testing)
3. Estimated survival time is more than 3 months in multiple myeloma,and Karnofsky Performance Status（KPS) score is more than 80.
4. No cytapheresis and cell separation contraindication.
5. Hemoglobin is more than 80 gram per litre.
6. The function of important organ was satisfied:(1)cardiac ultrasound indicated that cardiac ejection fractions is more than 50%（EF≥50%）, and the electrocardiogram showed no obvious abnormality;(2)Blood oxygen saturation is more than 90%（SpO2≥90%）;(3)Creatinine（Cr） is less than 2.5 times the upper limit of normal;(4)Alanine transaminase（ALT）and glutamic-oxalacetic transaminase（AST）is less than 3 times the upper limit of normal,and total bilirubin is less than 2 milligram per deciliter(TBil≤2.0mg/dL).
7. After discussion by the expert group, the patient's condition was analyzed and combined with the general physical condition of the patient, the benefit of participating in the clinical trial was greater than the risk.
8. Volunteered for this clinical trail and signed a consent form .
9. Currently, chemotherapy and approved targeted therapies are ineffective for the patients.Or patients cannot tolerate current chemotherapy.

Exclusion Criteria:

1. Active other disease and cannot control after treatment.
2. Patients with actively infection of Hepatitis B Virus (HBV) or Hepatitis C Virus (HCV).
3. Severe psychiatric disorder or other disease in central nervous system.
4. Patients are infected with fungus,bacteria or virus,and are difficult to control after treatment.
5. Patients with infection of HIV .
6. Pregnant or lactating women.
7. Patients who have Graft-Versus-Host Disease (GVHD) should receive systemic administration of immunosuppressive agents.
8. Patients have received other genetic therapy products.
9. Patients who have received systemic administration of glucocorticoid agents in one week before CART therapy.
10. Any situation may do harm to the subjects or interfere the results.
11. Have had Prolonged QT interval or severe heart disease in the past.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Adverse events that Are related to treatment | 2 years
  Determine the toxicity profile of the CD38/CD33/CD56/CD123/CD117/CD133/CD34/ Mucl-targeted CAR-T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0

SECONDARY OUTCOMES:
Estimate 2 year overall survival(OS) after infusion of CD38/CD33/CD56/CD123/ CD117/CD133/CD34/Mucl-CART and sequential treatment | 2 years
  To estimate 2 year overall survival(OS) after CD38/CD33/CD56/CD123/CD117/CD133/ CD34/Mucl-CART infusion and sequential treatment with Relapsed/Refractory AML
Estimate 2 year relapse rate after infusion of CD38/CD33/CD56/CD123/CD117/CD133/ CD34/Mucl-CART and sequential treatment | 2 years
  To estimate 2 year relapse rate after CD38/CD33/CD56/CD123/CD117/CD133/CD34/ Mucl-CART infusion and sequential treatment with Relapsed/Refractory AML
Estimate 2 year progression free survival after CD117/CD133/CD34/ Mucl-CART and sequential treatment | 2 years
  To estimate 2 year progression free survival after CD38/CD33/CD56/CD123/CD117/ CD133/CD34/Mucl-CART infusion and sequential treatment with Relapsed/Refractory AML

CONTACTS AND LOCATIONS:
Overall Officials: Yanjie He, Principal Investigator — Zhujiang Hospital
Locations (1):
- Southern Medical University Zhujiang Hospital, Guangdong, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided